CLINICAL TRIAL: NCT06900491
Title: Development of a Regional Irritable Bowel Syndrome Cohort
Brief Title: Irritable Bowel Syndrome Regional Cohort
Acronym: COSII
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0143/OB; IDRCB : 2024-A02023-44 (Other: ANSM)
Record Dates: First submitted 2025-03-14; First posted 2025-03-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The aim of setting up this biological collection is to be able to analyse the microbiota and the metabolites produced longitudinally. There will be a unique collection of saddles
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with irritable bowel syndrome: Patients with irritable bowel syndrome according to the Rome criteria in force at the time of inclusion (IV in 2024, V expected in 2025)
  Interventions: Other: self-questionnaires; Other: unique collection of saddles

INTERVENTIONS:
Other: self-questionnaires — Patients will fill in these self-questionnaires on a tablet or on paper, depending on the availability of tablets in the centres, before and after consulting the doctor. These questionnaires assess the severity of the disease and quality of life.
Other: unique collection of saddles — Stool samples will be taken at each visit, i.e. approximately every 6 months for patients

SUMMARY:
Setting up a regional (multicentre), longitudinal cohort of people suffering from irritable bowel syndrome followed up in consultation to study the natural history of the disease and its prognosis.

DETAILED DESCRIPTION:
The strategy of this project is to develop a regional cohort of patients suffering from irritable bowel syndrome, in order to offer harmonised phenotyping, longitudinal follow-up and the study of clinical and biological factors associated with the development of the disease and its treatment.

To achieve this, the study plans to prospectively collect a complete phenotyping of patients suffering from IBS and followed up in consultation in the participating centres (questioning, questionnaires, physiological explorations and results of complementary examinations), with follow-up of the course of the disease and which will be supplemented by stool samples for analyses of the microbiota and metabolites.

The study aims to include all patients seen prospectively in the centres over a period of 3 years and to include as many stool samples as possible during follow-up visits. This should make it possible to include a total of 600 patients. This number will be sufficient to identify subgroups of patients with similar clinical or biological characteristics of reasonable size (at least 50 to 100 subjects each) and then compare their prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient
* Normal laboratory work-up as part of routine care (CBC, CRP)
* Over 18 years of age
* Patient affiliated to a social security scheme
* Person who has read and understood the information letter and does not object to taking part in the study

Exclusion Criteria:

* Patient suffering from an organic digestive pathology (chronic inflammatory bowel disease, microscopic colitis when endoscopy has been performed because deemed necessary, digestive cancer, coeliac disease) or major digestive surgery (excluding appendectomy and cholecystectomy).
* Patient refusal
* Patient does not speak or understand French
* A pregnant woman or a woman in labour or breastfeeding
* Person deprived of liberty by an administrative or judicial decision or person placed under court protection / sub- guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients suffering from IBS referred to our centres for treatment will be consecutively included in the cohort. Patients will be selected by all hepato-gastroenterologists.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2030-09-04 (Estimated); Study Completion 2030-09-04 (Estimated)

PRIMARY OUTCOMES:
Clinical prognostic factors for the disease (use of recreational substances) | Visit V0 (inclusion)
  Assessing the use of amphetamines, LSD, cannabis, marijuana, heroin, cocaine, ecstasy, ketamine and methadone
Clinical prognostic factors for the disease (clinical history) | Visit V0 (inclusion)
  Assessment of antecedents: appendectomy, cholecystectomy, digestive surgery, diabetes and co-morbidities: fibromyalgia, chronic fatigue syndrome, migraine, hypermobility syndrome or Ehlers Danlos, eating disorders, ARFID, endometriosis or adenomyosis, insomnia and sleep disorders.
Clinical prognostic factors for the disease (use of treatment) | Visit V0 (inclusion)
  Assessment of the patient's use of probiotics, antispasmodics, analgesics, morphine, transit slowers, laxatives, psychiatric treatments, diets and alternative treatments.
Clinical prognostic factors for the disease (HAD score) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Assessment of stress (HAD score : Hospital Anxiety and depression scale (score ranging from 0 to 21)
Evaluation of validated questionnaires (SCOFF-F questionnaire) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Evaluation of patient responses to the SCOFF-F questionnaire (medical interview on weight loss or gain),
Evaluation of validated questionnaires (NIAS questionnaire (ARFID)) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Evaluation of patient responses to the NIAS questionnaire (ARFID) (Evaluation of food intake restriction or avoidance disorder: clinical characteristics characteristics ),
Evaluation of validated questionnaires (Francis score) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Evaluation of patient responses to the Francis score (Assessment of symptoms associated with irritable bowel syndrome (score from 0 to 500), the higher the score, the more severe the disease),
Evaluation of validated questionnaires (GIQLI score) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Evaluation of patient responses to the GIQLI score (Digestive quality of life score comprising 36 items covering symptoms, physical status, emotions, social problems and the effect of medical treatments. The score ranges from 0 to 144; the higher the score, the better the quality of life).
Evaluation of validated questionnaires (Fear of food questionnaire) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Evaluation of patient responses to the Fear of food questionnaire (The Fear of Food Questionnaire (FFQ) is an 18-item self-report questionnaire that measures fear, avoidance of food, as well as life interference and loss of pleasure from eating. Items are rated on a Likert scale ranging from 0 (not at all) to 5 (absolutely). Qualitative score ranges are 0-15 (minimal), 16-30 (mild), 31-45 (moderate), and 46-90 (severe))
Evaluation of validated questionnaires (EQ-5D-5L score) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Evaluation of patient responses to the EQ-5D-5L score (The EQ-5D-5L1 questionnaire is a European quality of life scale. The first part contains questions known as the 'EQ-5D descriptive system', supplemented by a visual analogue scale known as the 'EQ-5D VAS'. It consists of a 20 cm, graduated from 0 to 100, on which the patient is asked to indicate how they rate their current state of health, with 0 being the worst possible state and 100 being the best. and 100 being the best.).
Clinical prognostic factors for the disease (medical interview) | Visit V0 (inclusion)
  Assessment of sexual or physical aggression (medical interview), post-infectious nature (medical interview)
Clinical prognostic factors for the disease (Food avoidance questionnaire/exclusion diet) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Assessment of link with diet (Food avoidance questionnaire/exclusion diet informations)
Evaluation of validated questionnaires (VSI Score) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  A standardized psychological questionnaire that assesses coping strategies, that is, how a person deals with stress. 15 items describe a possible reaction to stress. For each of the 15 items, the person indicates to what extent the described reaction corresponds to them when they are stressed (in the face of pain, constipation, bloating, or an urgent need to go to the toilet). Six rating scales are used, ranging from: 1 strongly agree, 2 somewhat agree, 3 slightly agree, 4 slightly disagree, 5 somewhat disagree, and 6 strongly disagree
Evaluation of validated questionnaires (PHQ15 Score) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Screening for somatic symptoms (frequent physical complaints). 15 items corresponding to a physical symptom. 3 levels of response: score 0 means no somatic symptoms, score 1 means mild somatic symptoms, and score 2 means severe somatic symptoms
Evaluation of validated questionnaires (CISS) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  This assessment evaluates an individual's cognitive and behavioral efforts to manage a situation perceived as stressful. Seven items, each worth 5 points, assess a single coping style (minimum score of 7 and maximum of 28). A low score indicates limited cognitive and behavioral effort in managing a situation perceived as stressful.

SECONDARY OUTCOMES:
Metabolomic analyses | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  Metabolomics by GC-MS and LC-MS, lipidomics, SCFAs, bile acids
analyses carried out on stool samples (metagenomic shotgun) | Visit V0 (inclusion), Visits at 6 , 12, 18, 24, 30 and 36 months
  metagenomic shotgun analysis of microbiota (composition of the microbiota)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - University Hospitol of Amiens, Amiens
  - CHU de CAEN, Caen
  - University Hospital of Lille, Lille
  - University Rouen Hospital, Rouen

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.